CLINICAL TRIAL: NCT01016821
Title: The Efficacy and Safety of Intravenous Oxycodone and Plasma Oxycodone Concentrations in Labour Pain
Brief Title: Oxycodone for Labor Pain - Pharmacokinetics (PK), Safety and Efficacy
Acronym: Oksiobs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Merja Kokki, PhD, Kuopio University Hospital, Department of Anaesthesiology and Intensive Care
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KUH5070213; 2009-013469-25 (Other: Eudra CT number)
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Labor Pain
Keywords: Oxycodone; Labour pain; Pregnancy; Pregnant women
MeSH Terms: conditions — Labor Pain | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxycodone, labour pain (Other)
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — Intravenous, 1 mg, 5 times, in every 5 minutes, duration of drug administration 25 minutes

SUMMARY:
Childbirth is one of the most painful events that a woman is likely to experience, and thus is a major concern for most parturient. Severe pain releases stress mediators and may thus compromise fetus well-being if placental perfusion is decreased. Epidural analgesia is the golden standard for the management of severe labor pain. However, it could not always be used both due the parturient related factors and the organizational reasons.However, the knowledge on safety and efficacy of oxycodone involving mother, fetus and newborn is limited.

Aim of the study is firstly, to evaluate the efficacy and safety of oxycodone in labor pain healthy parturients. Secondly, to measure parturient's blood oxycodone concentration during labour and fetal concentration from placental umbilical vein and artery right after birth.

ELIGIBILITY:
Inclusion Criteria:

* Labouring healthy women
* Early labour
* Age 18-45 years

Exclusion Criteria:

* Sleep apnea or other central deficit affecting breathing
* Pulmonary insufficiency
* Liver of kidney insufficiency
* Use of mono amine oxidase medication
* Thyroid, pituitary insufficiency
* Paralytic ileus
* Other contraindication specified by the investigator

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The efficacy and safety of oxycodone in labor pain | 24 hours

SECONDARY OUTCOMES:
The parturient's blood oxycodone concentration during labour and fetal concentration from placental umbilical vein and artery right after birth | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Merja Kokki, PhD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland